CLINICAL TRIAL: NCT03906994
Title: Treating Amblyopia in Adults With Interactive Video Games
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original study PI left institution and the new PI elected not to proceed with the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erick D. Bothun, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000212
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with Amblyopia (Experimental): Adult amblyopia subjects will play the video game Mario Kart Wii
  Interventions: Other: Video game Mario Kart Wii

INTERVENTIONS:
Other: Video game Mario Kart Wii — Subjects will place a patch over the better-seeing eye and play the video game Mario Kart Wii for a total of 40 hours over a 1 month perior

SUMMARY:
Researchers are trying to determine whether interactive video game play, while wearing a patch over better-seeing eye, will improve subject reduced vision (amblyopia).

DETAILED DESCRIPTION:
The purpose of this research is to determine whether amblyopia (reduced vision in one eye) in adults can be improved using interactive video game play.

Study participation involves playing the video game Mario KartTM (provided by the study), while wearing a patch over their better-seeing eye. Participants are asked to play the game for a total of 40 hours over a one-month period.

The primary outcome measure will be LogMAR visual acuity measured 1 month after initiating game play.

ELIGIBILITY:
Inclusion Criteria:

* Aged >17 years old
* Refraction within past year and wearing updated glasses or contact lenses
* Diagnosis of strabismic, anisometropic or combined amblyopia (> 2 lines inter-ocular difference)
* Stable visual acuity as defined as <1 LogMAR change over 2 visits 8 weeks apart, or wearing glasses for at least 16 weeks

Exclusion Criteria:

* Monovision and unwilling to wear corrective glasses
* Allergy to adhesive bandages
* Women who are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity | Baseline, one month
  measured using the LogMAR (Logarithm of the Minimum Angle of Resolution) chart comprised of rows of letters to estimate visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Erick Bothun, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials